CLINICAL TRIAL: NCT04222582
Title: The Neural, Behavioural, and Cognitive Outcomes of Transcranial Direct Current Stimulation (tDCS) for Persistent Auditory Verbal Hallucinations in Schizophrenia
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Persistent Auditory Verbal Hallucinations in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Collaborators: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Verner Knott, Senior Scientist, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017020
Record Dates: First submitted 2019-04-15; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Auditory Hallucination, Verbal
Keywords: Schizophrenia; Transcranial direct current stimulation (tDCS); Schizoaffective disorder; EEG; Brain imaging; Cognition
MeSH Terms: conditions — Hallucinations; Schizophrenia; Psychotic Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active tDCS (Active Comparator): Administration of a 2 milliamp (mA) current delivered via two scalp electrodes for 20 minutes (ramp-in + ramp-out periods, 30s total) 2 times per day for 5 consecutive days, >3 hour interval between sessions, for a total of 10 tDCS sessions.
  tDCS will be administered with a constant current regulator (NeuroConn DC-Stimulator Plus®, Germany) using 2 saline-soaked sponge electrodes applied over the scalp. Using the 10-20 international EEG system for tDCS electrode placement, the anode will be positioned midway between F3 and Fp1 (left DLPFC) and the cathode midway between T3 and P3 (left TPJ).
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): Administration of 2mA tDCS for 30 seconds followed by 19.5 minutes of no current via two scalp electrodes for 20 min (2X/day for 5 consecutive days) with >3 hours interval between sessions, for a total of 10 tDCS sessions.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Open-label Active tDCS (Other): Subjects who have received sham tDCS will be given the option to subsequently receive 10 sessions of open-label active tDCS (2X/day for 5 consecutive days) with >3 hours interval between sessions, for a total of 10 tDCS sessions.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Healthy Control (No Intervention): Healthy volunteers will complete the same questionnaires, EEG recording procedures, and neuroimaging scans as the schizophrenia patient group, but will not undergo tDCS.

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation (tDCS) is a non-invasive form of brain stimulation which uses a weak current (2mA direct current) to temporarily excite or inhibit underlying brain regions with small electrodes placed on the scalp.
  Arms: Active tDCS; Open-label Active tDCS; Sham tDCS

SUMMARY:
Many individuals with schizophrenia struggle with auditory verbal hallucinations (AVHs). In some cases, these AVHs can be resistant to medication treatment. Previous research has found that transcranial direct current stimulation (tDCS) can be helpful in treating symptoms in individuals with other psychiatric disorders, such as depression. This study will assess if tDCS is effective in treating AVHs in individuals with schizophrenia. tDCS is a non-invasive form of brain stimulation which uses a weak current to temporarily excite or inhibit underlying cortical regions with small electrodes placed on the scalp. tDCS has been found to improve mental processes, including attention and memory function. In addition to examining the effect of tDCS on AVHs, this study will assess the effects of tDCS on mood as well as brain electrical activity with electroencephalogram (EEG) recordings. As an additional component, participants will be invited to participate in neuroimaging. Using magnetic resonance imaging (MRI), brain activity and structure will be examined before and after tDCS. tDCS will be administered twice daily for 5 consecutive days for a total of 10 sessions. These study findings will contribute to the understanding of the impact of tDCS on AVHs, and will also increase knowledge of sound and memory/cognitive processing in individuals with schizophrenia.

ELIGIBILITY:
Patients - Inclusion Criteria:

* Primary diagnosis of schizophrenia or schizoaffective disorder
* Clinically stable (discretion of psychiatrist)
* Consistent history of AVHs over the course of illness
* >3 AVHs per week
* Positive and Negative Syndrome Scale (PANSS) score of >3
* Primary medications limited to one of the atypical antipsychotics (medications stabilized for 4 weeks prior to enrollment)

Patients - Exclusion Criteria:

* Experiencing an acute psychotic episode
* Current drug/alcohol dependence
* Significant medical illness & mental retardation/learning disability
* Extra-pyramidal symptoms resulting in disordered movement
* Abnormal audiometric assessment (thresholds for pure tones >25 dB)
* History of significant neurological issues & head injuries/concussions resulting in loss of consciousness for >5 minutes

Healthy Controls - Inclusion Criteria:

* In good physical health
* No history of serious mental health issues

Healthy Controls - Exclusion Criteria:

* Personal history of psychiatric disorder
* Family history of schizophrenia in first degree relatives & history of mental health issues in first degree relatives that required extensive treatment or hospitalization
* Current/history of substance abuse
* Significant medical illness
* Extra-pyramidal symptoms resulting in movement disorder
* Abnormal audiometric assessment (thresholds for pure tones >25 dB)
* Significant neurological issues & head injuries/concussions resulting in loss of consciousness for >5 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in auditory hallucination severity measured by the Psychotic Symptom Rating Scale (PSYRATS) | Baseline, after 2nd tDCS session on days 1, 3, and 5, and follow-up (within a week of completing tDCS)
  The PSYRATS is a multidimensional measure of auditory hallucinations, including 11 items rated on five-point (0-4) scales (total score range 0-44). Symptoms are rated over the last week, with higher scores reflecting more severe symptoms. The dimensions assessed are frequency, duration, location, loudness, beliefs about origin, negative content, intensity of negative content, amount of distress, intensity of distress, disruption of life and control.

SECONDARY OUTCOMES:
Change in Voice Power Differential Scale (VPDS) Scores | 3 weeks (baseline to follow-up)
  The Voice Power Differential Scale (VPDS) is a 7-item scale used to measure the perceived power differences between the voice and the voice hearer. Each item is rated on a five-point scale (1-5), with higher scores indicating greater power differential in favour of the voices, with total scores ranging from 7-35.
Change in Beliefs about Voices Questionnaire-Revised (BAVQ-R) Scores | 3 weeks (baseline to follow-up)
  The BAVQ-R is a 35-item questionnaire assessing people's beliefs about auditory hallucinations, and their emotional and behavioural reactions to them. All responses are rated on a 4-point scale: disagree (0); unsure (1); agree slightly (2); agree strongly (3), the measure thus assesses degree of endorsement of items. The scale consists of five subscales: malevolence (score range 0-18), benevolence (0-18), omnipotence (0-18), resistance (0-27), and engagement (0-24).
Change in Voices Acceptance and Action Scale (VAAS) Scores | 3 weeks (baseline to follow-up)
  The VAAS was developed to assess acceptance-based or action-based beliefs in response to auditory verbal hallucinations, in general and specifically to command hallucinations. This 31-item scale is divided into section A (i.e., 12 item stand-alone scale for general auditory hallucinations) and section B, referring specifically to command hallucinations. The participant is asked to rate their opinion from 1 'Strongly Disagree' to 5 'Strongly Agree', with higher scores meaning higher levels of acceptance and perception of acting according to one's valued life directions. Section A scores can range from 12-60, while section B scores can range from 19-95.
Change in Electroencephalography (EEG) - Resting-State Alpha Power | 3 weeks (baseline to follow-up)
  Changes in resting-state EEG power in alpha band. Resting-state recordings completed in both eyes-closed and eyes-open conditions, 5 minutes each.
Change in Electroencephalography (EEG) - Resting-State Beta Power | 3 weeks (baseline to follow-up)
  Changes in resting-state EEG power in beta band. Resting-state recordings completed in both eyes-closed and eyes-open conditions, 5 minutes each.
Change in Electroencephalography (EEG) - Resting-State Delta Power | 3 weeks (baseline to follow-up)
  Changes in resting-state EEG power in delta band. Resting-state recordings completed in both eyes-closed and eyes-open conditions, 5 minutes each.
Change in Electroencephalography (EEG) - Resting-State Theta Power | 3 weeks (baseline to follow-up)
  Changes in resting-state EEG power in theta band. Resting-state recordings completed in both eyes-closed and eyes-open conditions, 5 minutes each.
Change in Electroencephalography (EEG) - Resting-State Gamma Power | 3 weeks (baseline to follow-up)
  Changes in resting-state EEG power in gamma band. Resting-state recordings completed in both eyes-closed and eyes-open conditions, 5 minutes each.
Change in Electroencephalography (EEG) - Mismatch Negativity (MMN) | 3 weeks (baseline to follow-up)
  Change in MMN peak amplitudes and latencies to non-speech (tonal) deviants and speech (syllabic) deviants during the multi-feature optimal MMN paradigm.
Change in Electroencephalography (EEG) - P50 | 3 weeks (baseline to follow-up)
  Change in T/C ratio (testing stimulus/conditioning stimulus) during paired click test.
  Change in T/C difference (testing stimulus - conditioning stimulus) during paired click test
Change in Brain Functional Magnetic Resonance Imaging (fMRI) - Resting-State | 3 weeks (baseline to follow-up)
  Changes in resting-state activity and connectivity within and between the auditory cortex and select regions of the default-mode network.
Change in Brain Functional Magnetic Resonance Imaging (fMRI) - Mismatch Negativity (tonal) | 3 weeks (baseline to follow-up)
  Changes in task-related activity and connectivity within and between the auditory cortex and select regions of the default-mode network .
Change in Brain Magnetic Resonance Spectroscopy (MRS) | 3 weeks (baseline to follow-up)
  Changes in glutamate/glutamine (Glu/Gln) concentrations in the auditory cortex.
Change in Cambridge Neuropsychological Test Automated Battery (CANTAB) Schizophrenia Battery | 3 weeks (baseline to follow-up)
  Changes in cognitive functioning abilities in core domains often affected in psychosis.
Change in Social Cognition - Social Attribution Task | 3 weeks (baseline to follow-up)
  Changes in social cognition/social inference abilities measured by a computerized social attribution task.

CONTACTS AND LOCATIONS:
Overall Officials: Verner Knott, PhD, C.Psych, Principal Investigator — University of Ottawa; Natalia Jaworska, PhD, Principal Investigator — University of Ottawa
Locations (1):
- Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No